CLINICAL TRIAL: NCT02680626
Title: Bilateral Transversus Abdominis Plane Block With or Without Magnesium for Total Abdominal Hysterectomy With or Without Salpingo-oophorectomy: a Randomized Controlled Trial
Brief Title: Bilateral Transversus Abdominis Plane Block With or Without Magnesium
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Pfannenstiel hysterectomies are now rarely performed so cannot recruit eligible patients
Sponsor: Dr. Anthony Ho (Other)
Responsible Party: Sponsor-Investigator, Dr. Anthony Ho, Professor, GFT, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAE-275-15
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium (Experimental): Participants in this arm will receive magnesium sulfate + ropivacaine in their bilateral transversus abdominis plane blocks
  Interventions: Drug: Magnesium Sulfate; Drug: Ropivacaine
- Non-magnesium (Active Comparator): Participants in this arm will receive saline + ropivacaine in their bilateral transversus abdominis plane blocks
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Magnesium Sulfate — Given via transversus abdominis plane block
  Other Names: Sulfamag, Epsom salt, Health Canada DIN: 02139499
  Arms: Magnesium
Drug: Ropivacaine — Given via transversus abdominis plane block
  Other Names: Naropin

SUMMARY:
Pain control after surgery is important for patient well-being and recovery. We are interested in determining whether we can improve the duration of action of a local anesthetic procedure (transversus abdominis plane block, or TAP block) by adding magnesium sulfate to local anesthetics given to patients after total abdominal hysterectomy with or without salpingo-oophorectomy.

DETAILED DESCRIPTION:
Total abdominal hysterectomy (TAH) with or without salpingo-oophorectomy is a commonly performed major surgical procedure that results in significant postoperative pain. Traditionally, this pain has been treated with a multimodal approach which includes opioids, often administered via a patient-controlled analgesia (PCA) pump. Common side effects of opioids include sedation, nausea, vomiting, constipation, and pruritus. Thus, to overcome such undesirable side effects, other approaches to pain management have been explored, including post-operative transversus abdominis plane (TAP) blocks. TAP blocks are a popular analgesia technique for abdominal surgery with an incision between the sixth thoracic (T10) vertebrae and the first lumbar (L1) vertebrae. The block involves infiltration of local anesthetic (LA) by an anesthesiologist under direct ultrasound guidance. The anesthetic is deposited into a plane between the internal oblique and transversus abdominis muscles, which contain thoracolumbar nerves that originate from the T6 to L1 spinal roots. These nerves supply sensation to the anterolateral abdominal wall, the area responsible for incision-related pain following TAH ± unilateral/bilateral salpingo-oophorectomy. TAP blocks are a low risk procedure with very rare side-effects including bowel or peritoneum perforation, and local anesthetic toxicity. Almost all anesthesiologists are familiar with performing such a block, which is routinely done under ultrasound guidance to minimize the risk of perforation. Previous studies demonstrate TAP block efficacy in various abdominal surgery including hysterectomy, colon resection, Caesarean section, retropubic prostatectomy, laparoscopic cholecystectomy, and open appendectomy. While TAP blocks have been shown to provide patients with a statistically significant increase in the time to first analgesic request, this mean delay is typically less than 3 hours. To overcome the limited duration of action, we are proposing the addition of magnesium as an adjunct to the LA solution infiltrated in the block. Other regional anesthesia techniques have trialed various adjuncts including epinephrine, dexamethasone, clonidine, and recently magnesium. The goal of using such adjuncts is to prolong and enhance analgesia, and potentially even decrease total LA required. Our study will investigate the use of magnesium as an adjunct to LA in bilateral TAP blocks to increase the duration of analgesia. Magnesium is the fourth most abundant cation in the body and the second most abundant intracellular cation after potassium. The minimum recommended daily intake of magnesium for adults is 0.25 mmol (6 mg)/kg body weight. Magnesium is a natural analgesic through antagonism of N-methyl-D-aspartate receptors. When added to LA, magnesium has been shown to improve the quality and duration of analgesia of neuraxial, femoral, and brachial plexus blocks. In fact, brachial plexus analgesia has been produced with magnesium sulfate (MgSO4) alone. Magnesium as an adjunct to TAP blocks has never been previously investigated in any setting, thus we propose a study to specifically investigate its potential effects in prolonging analgesia in patients undergoing elective TAH ± unilateral or bilateral salpingo-oophorectomy. We hypothesize that the quality and duration of analgesia can be improved by adding a moderate amount of MgSO4 to the local anesthetic used in the TAP blocks.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) rating I-III
* Age 18-75 years old
* Female
* Undergoing elective total abdominal hysterectomy (TAH) with or without uni/bilateral salpingo-oophorectomy (BSO) under general anesthesia with a Pfannenstiel incision
* Admitted to hospital postoperatively (inpatients)
* Competent to provide informed consent

Exclusion Criteria:

* Emergency TAH ± BSO
* ASA IV-V
* Allergy or sensitivity to study-related medications
* Taking any medications that are contraindicated for the use of any of our study drugs
* Midline incision
* Other regional anesthesia technique (e.g. epidural)
* Morbidly Obese (BMI > 40)
* Incompetent to provide informed consent
* eGFR < 50
* Impaired liver function (INR > 1.5)
* Pre-existing chronic pain condition requiring chronic opioid use
* Significant co-existing cardiovascular disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-01; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Time to first dose of post-operative opioid | First occurrence during hospitalization (up to 24 hours postoperatively)
  Investigators will note the time lapsed between end of surgery (when TAP block administered) and the first request for additional analgesia (given using patient controlled analgesia pumps, as is standard of care at our institution).
Cumulative opioid consumption | Cumulative dose consumed at 2, 4, 6, 8, and 25 hours after receiving TAP blocks
  Investigators will record the total amount of opioid consumed between receiving the TAP block and 24 hours later.

SECONDARY OUTCOMES:
Pain score | 2, 4, 6, 8, and 24 hours after receiving TAP block
  Visual analog scales will be used to assess pain at rest and upon coughing in patients at various time points after receiving the TAP block after surgery.
Time to post-anesthetic care unit discharge | First occurrence during the initial 24 hours after surgery
  Investigators will note the time lapsed between a patient receiving their TAP block and when she is discharged from the PACU.
Nausea score | 2, 4, 6, 8, and 24 hours after receiving TAP block
  Nausea will be rated from 0 (none) to 3 (vomiting) at various time points after receiving TAP block
Pruritis score | 2, 4, 6, 8, and 24 hours after receiving TAP block
  Pruritis will be rated from 0 (none) to 3 (severe) at various time points after receiving TAP blocks.
Sensory block | 30 minutes after arrival into the post-anesthetic care unit, and at 2, 4, 6, and 8 hours after receiving TAP blocks
  Ice will be placed on each side of the abdomen and on the upper arm. The participant will be asked if she can feel the ice on her abdomen, and if it feels similar to that on her upper arm.
Patient satisfaction | At 24 hours after receiving TAP blocks
  Participants will be asked to rate their satisfaction from 1 (poor) to 4 (excellent)
Quality of Recovery score | At 24 hours after receiving TAP blocks
  Participants will be asked to fill out this 9-part survey, which consists of rating 9 statements related to recovery from anesthetic and surgery on a scale from 0 (not at all) to 2 (most of the time)
Side effects | At 24 hours after receiving TAP blocks
  Participants will be asked whether they experienced any side effects during the 24 hours between receiving TAP block and end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Ho, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gasanova I, Grant E, Way M, Rosero EB, Joshi GP. Ultrasound-guided transversus abdominal plane block with multimodal analgesia for pain management after total abdominal hysterectomy. Arch Gynecol Obstet. 2013 Jul;288(1):105-11. doi: 10.1007/s00404-012-2698-3. Epub 2013 Jan 6. PMID 23291970
- [Background] Siddiqui MR, Sajid MS, Uncles DR, Cheek L, Baig MK. A meta-analysis on the clinical effectiveness of transversus abdominis plane block. J Clin Anesth. 2011 Feb;23(1):7-14. doi: 10.1016/j.jclinane.2010.05.008. PMID 21296242
- [Background] Griffiths JD, Le NV, Grant S, Bjorksten A, Hebbard P, Royse C. Symptomatic local anaesthetic toxicity and plasma ropivacaine concentrations after transversus abdominis plane block for Caesarean section. Br J Anaesth. 2013 Jun;110(6):996-1000. doi: 10.1093/bja/aet015. Epub 2013 Mar 1. PMID 23454825
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] O'Donnell BD, McDonnell JG, McShane AJ. The transversus abdominis plane (TAP) block in open retropubic prostatectomy. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):91. doi: 10.1016/j.rapm.2005.10.006. No abstract available. PMID 16418039
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789
- [Background] Niraj G, Searle A, Mathews M, Misra V, Baban M, Kiani S, Wong M. Analgesic efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing open appendicectomy. Br J Anaesth. 2009 Oct;103(4):601-5. doi: 10.1093/bja/aep175. Epub 2009 Jun 26. PMID 19561014
- [Background] Bonnet F, Berger J, Aveline C. Transversus abdominis plane block: what is its role in postoperative analgesia? Br J Anaesth. 2009 Oct;103(4):468-70. doi: 10.1093/bja/aep243. No abstract available. PMID 19749115
- [Background] Schlingmann KP, Konrad M, Seyberth HW. Genetics of hereditary disorders of magnesium homeostasis. Pediatr Nephrol. 2004 Jan;19(1):13-25. doi: 10.1007/s00467-003-1293-z. Epub 2003 Nov 22. PMID 14634861
- [Background] Fawcett WJ, Haxby EJ, Male DA. Magnesium: physiology and pharmacology. Br J Anaesth. 1999 Aug;83(2):302-20. doi: 10.1093/bja/83.2.302. PMID 10618948
- [Background] James MF. Clinical use of magnesium infusions in anesthesia. Anesth Analg. 1992 Jan;74(1):129-36. doi: 10.1213/00000539-199201000-00021. No abstract available. PMID 1734773
- [Background] El-Shamaa HA, Ibrahim M, Eldesuky HI. Magnesium sulfate in femoral nerve block, does postoperative analgesia differ? A comparative study. Egypt Journal of Anaesthesia 30(2): 169-73, 2013
- [Background] Lee AR, Yi HW, Chung IS, Ko JS, Ahn HJ, Gwak MS, Choi DH, Choi SJ. Magnesium added to bupivacaine prolongs the duration of analgesia after interscalene nerve block. Can J Anaesth. 2012 Jan;59(1):21-7. doi: 10.1007/s12630-011-9604-5. Epub 2011 Oct 20. PMID 22012543
- [Background] Gunduz A, Bilir A, Gulec S. Magnesium added to prilocaine prolongs the duration of axillary plexus block. Reg Anesth Pain Med. 2006 May-Jun;31(3):233-6. doi: 10.1016/j.rapm.2006.03.001. PMID 16701189
- [Background] Abdelfatah AM, Elshaer AN. The effect of adding magnesium sulfate to lidocaine in an interscalene plexus block for shoulder arthroscopic acromioplasty. Ain-Shams Journal of Anesthesiology 7(1): 59-64, 2014.
- [Background] Yousef GT, Ibrahim TH, Khder A, Ibrahim M. Enhancement of ropivacaine caudal analgesia using dexamethasone or magnesium in children undergoing inguinal hernia repair. Anesth Essays Res. 2014 Jan-Apr;8(1):13-9. doi: 10.4103/0259-1162.128895. PMID 25886097
- [Background] Goyal P, Jaiswal R, Hooda S, Hoyal R, Lal J. Role of magnesium sulphate for brachial plexus analgesia. Internet Journal of Anesthesiology. 21(1): 1-6, 2008.